CLINICAL TRIAL: NCT06343428
Title: Definition of a Multiparametric Prognostic and Predictive System of Classification of NET G3 Patients: an observAtional, Prospective Analysis of the Correlation Between Functional Imaging and Clinical Outcome (TAPIOCA)
Brief Title: Definition of a Multiparametric Prognostic and Predictive System of Classification of NET G3 Patients
Acronym: TAPIOCA
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1519
Record Dates: First submitted 2024-03-18; First posted 2024-04-02 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-03

CONDITIONS: Neuroendocrine Neoplasm
Keywords: High-grade neuroendocrine neoplasm; prognostic factor; predictive factor
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample, tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NET G3 patients: Histological diagnosis of well-differentiated neuroendocrine tumor G3 performed or reviewed by a NEN-dedicated pathologist.

SUMMARY:
The 2017 World Health Organization (WHO) introduced a new category of high-grade, well-differentiated neuroendocrine neoplasms (NENs) that called neuroendocrine tumors (NETs) G3 in pancreatic NENs classification and, then, in 2019, for all gastro-entero-pancreatic (GEP) tract NENs.

The new classification made it possible to separate NETs G3 from high-grade, poorly-differentiated, NENs that are called neuroendocrine carcinomas (NECs).

However, in clinical practice, we observed that several clinical, pathological and radiological differences are arising among NET G3 patients, suggesting that a multiparametric definition of NET G3 is needed.

DETAILED DESCRIPTION:
High-grade neuroendocrine neoplasms (NENs) represent the poorest prognosis category within NENs. During the years, the prognostic differences among the subgroups led to identify at least two subcategories of high-grade NENs, according the morphologic features of the two subtypes.

Indeed, the 2017 World Health Organization (WHO) introduced a new category of high-grade, well-differentiated NENs that called neuroendocrine tumors (NETs) G3 for pancreatic NENs and, then, in 2019, for all gastro-entero-pancreatic (GEP) tract NENs, allowing to separate NET G3 from the other high-grade, poorly-differentiated, NENs, so called neuroendocrine carcinomas (NECs).

However, since the new-category has been introduced, NET G3 category seemed to be more heterogeneous than presumed. Indeed, clinical, pathological and radiological features seemed to identify different prognostic subcategories of NET G3. We recently performed a retrospective analysis on a small pool of 48 NET G3 patients, correlating the clinical outcomes with these different features. The results of our study seemed to suggest prognostic and predictive factors that deserve to be prospectively explored to better understand this pathology and that might to be part of NET G3 multiparametric classification system. Based on the results of our retrospective analysis, we underlined the importance of a systematic and well-designed collection of high-quality data in order to improve our knowledge on this topic.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of well-differentiated neuroendocrine tumor G3 performed or reviewed by a NEN-dedicated pathologist. In case of "late-NET G3" (see Patients and Methods), a NEN-dedicated pathologist will perform a pathologic review of the previous NET G1/2, too, unless a NEN-dedicated pathologist has already done and except for diagnoses performed in a NEN-referral Center.
* Age > 18 years
* Signed written informed consent
* Available tumor tissue (formalin-fixed paraffin-embedded, FFPE) (preferably within 6 months). If the tumor contained in FFPE tissue block cannot be provided in total, sections from this block should be provided that are freshly cut. Preferably, 25 slides should be provided (minimum of 15 slides). If tumor tissue is not available, patients should be willing to undergone to a new biopsy.
* late-NET G3 patients that will come to our Institute at the moment of NET G3 diagnosis will be enrolled only if they performed 68 Gallium-DOTATOC positron emission tomography (PET)/CT and 18 fluorodeoxyglucose (FDG)-PET/CT for the previous NET G1/2. The previous functional imaging performed during the NET G1/2 history shall be available for the review by our specialist in nuclear medicine.

Exclusion Criteria:

* Diagnosis of well-differentiated NET G1/2 or poorly-differentiated NEC
* Diagnosis of mixed neuroendocrine non-neuroendocrine neoplasms (MiNENs) in which a NET G3 as neuroendocrine component
* Cytological diagnosis of NET G3 or not availability of tumor tissue for pathological analysis
* Concurrent neoplastic disease (e.g. advanced breast or prostatic cancer in hormonal treatment, hematologic diseases)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: NET G3 patients managed at IEO. Histological diagnosis of well-differentiated neuroendocrine tumor G3 performed or reviewed by a NEN-dedicated pathologist. In case of "late-NET G3" a NEN-dedicated pathologist will perform a pathologic review of the previous NET G1/2, too, unless a NEN-dedicated pathologist has already done and except for diagnoses performed in a NEN-referral Center.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-07-19 (Actual); Primary Completion 2024-07-19 (Estimated); Study Completion 2026-07-19 (Estimated)

PRIMARY OUTCOMES:
Immunohistochemical characteristics analysis | 3 years
  Analysis of the morphology Analysis of proliferation index Ki-67 Analysis of Ki-67 expression (as hotspot or a diffuse expression on the sample) Analysis of Synaptophysin, and chromogranin expression

SECONDARY OUTCOMES:
Review of the functional imaging | 3 years
  Analysis of homogeneity or inhomogeneity of radiotracer distribution Analysis of the concordance/discordance between functional imaging. For "late-NET G3", the specialist in nuclear medicine will review both functional imaging (before and after NET G3 diagnosis)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Spada, MD, Principal Investigator — Istituto Europeo di Oncologia
Locations (1):
- European Institute of Oncology, Milan, Italy

IPD SHARING:
Plan to Share IPD: No